CLINICAL TRIAL: NCT03705676
Title: Unraveling the Puzzle of Back Pain Chronicity: an Integrative Perspective on Sensorimotor Control and Maladaptive Cognitive Processes
Brief Title: Unraveling Back Pain Chronicity: an EMG and EEG Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016/0186
Record Dates: First submitted 2018-09-05; First posted 2018-10-15 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
Keywords: Sensorimotor control; Event-related potentials; Cortical movement preparation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Each participant will perform both experimental conditions spread out over 2 test days in a randomized order. Between 2 test days a minimum of 5 days has to be present in order to ensure full recuperation from test day 1. Half of the participants will receive the control condition on test day 1 and the fear condition on day 2, the other half vice versa.
Who Masked: Outcomes Assessor
Masking Description: Participants are aware that electrocutaneous stimulation might occur during the fear condition and never during the control condition. This is of paramount importance, as the expectancy of a painful stimulus is the main difference between both conditions.
  The researcher that will perform the EMG-analysis, i.e. onset determination of the various muscles that were measured, will be blinded for participant, condition and muscle during that process. EEG-data does not have to be blinded as data processing is computer based and not subjectable to subjective bias of a researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy controls - control condition (Active Comparator): Assesses EMG and EEG activity of healthy controls during a rapid arm task after a warning and go cue. No painful stimuli are administered, only non-painful vibrotactile stimuli.
  Interventions: Behavioral: Rapid Arm Movements; Device: Vibrotactile stimulus
- Healthy controls - fear condition (Experimental): Assesses EMG and EEG activity of healthy controls during a rapid arm task after a warning and go cue. Half of the trials are no threat trials, the other half are threat trials. A painful stimulus is administered during arm movement in 25% of the threat trials in order to evoke anticipation of pain during the 75% other threat trials.
  Interventions: Behavioral: Rapid Arm Movements; Device: Unpleasant stimulus; Device: Vibrotactile stimulus
- RLBP - control condition (Active Comparator): Assesses EMG and EEG activity of RLBP subjects during a rapid arm task after a warning and go cue. No painful stimuli are administered, only non-painful vibrotactile stimuli.
  Interventions: Behavioral: Rapid Arm Movements; Device: Vibrotactile stimulus
- RLBP - fear condition (Experimental): Assesses EMG and EEG activity of RLBP subjects during a rapid arm task after a warning and go cue. Half of the trials are no threat trials, the other half are threat trials. A painful stimulus is administered during arm movement in 25% of the threat trials in order to evoke anticipation of pain during the 75% other threat trials.
  Interventions: Behavioral: Rapid Arm Movements; Device: Unpleasant stimulus; Device: Vibrotactile stimulus
- CLBP - control condition (Active Comparator): Assesses EMG and EEG activity of CLBP subjects during a rapid arm task after a warning and go cue. No painful stimuli are administered, only non-painful vibrotactile stimuli.
  Interventions: Behavioral: Rapid Arm Movements; Device: Vibrotactile stimulus
- CLBP - fear condition (Experimental): Assesses EMG and EEG activity of CLBP subjects during a rapid arm task after a warning and go cue. Half of the trials are no threat trials, the other half are threat trials. A painful stimulus is administered during arm movement in 25% of the threat trials in order to evoke anticipation of pain during the 75% other threat trials.
  Interventions: Behavioral: Rapid Arm Movements; Device: Unpleasant stimulus; Device: Vibrotactile stimulus

INTERVENTIONS:
Behavioral: Rapid Arm Movements — 240 trials of RAM in either a forward (50%) or backward (50%) shoulder flexion direction and back to neutral as fast as possible, with maintaining extension in the elbow. Visual cues (arrows) indicated the movement direction.
Device: Unpleasant stimulus — An unpleasant, but harmless, electrocutaneous stimulus is administered to the low back region in 25% of the threat trials during the fear condition. Due to a conditioning phase before testing, participants know to expect this stimulus after the presentation of a warning cue related to the fear trials (either pink or blue dot dependent on randomization).
  Other Names: Electrocutaneous stimulus
  Arms: CLBP - fear condition; Healthy controls - fear condition; RLBP - fear condition
Device: Vibrotactile stimulus — In all trials, during the presentation of the warning cue, a vibrotactile stimulus is administered to the low back region. This stimulus is used to evoke somatosensory evoked potentials (SEP) measured with EEG during the movement-preparation phase.

SUMMARY:
This study aims at examining the influence of both threat of experimentally induced pain and clinical low back pain (LBP) on trunk motor control on the one hand and brain activity related to movement preparation on the other hand. Therefore, 3 groups are studied: healthy controls, people with recurrent LBP, and people with chronic LBP. A comparison in electromyography (EMG) of the trunk muscles and electroencephalography (EEG) activity between the 3 groups will be made in 2 conditions: a control condition without experimental pain on 1 test day, and a fear condition with experimental pain on another test day. In both conditions a motor control task will be performed and muscle and brain activity will be measured during each motor control task.

It is hypothesised that motor control will be different between the 3 groups in both conditions, i.e. delayed trunk muscle onset in LBP groups compared with controls. With regards to the brain activity, it is expected that preparation for movement will also be delayed in the LBP groups. Furthermore, it is expected that the fear condition will entail differences in both EMG and EEG within each group.

DETAILED DESCRIPTION:
March 2017 - April 2018. 30 healthy participants, 30 recurrent and 30 chronic LBP patients all aged 18-45 and of both genders were tested for 2 conditions on 2 separate days, i.e. a control condition (C) on 1 test day; a fear (F) condition consisting out of threat (T) and no threat trials (NT) on another test day. The order of test days was randomized.

1 block of 240 rapid arm movements (RAM) with the dominant arm was performed per condition, while electroencephalography (EEG) of the brain and surface electromyography (sEMG) of the Internal Oblique/Transversus Abdominis, External Oblique, Multifidus and Iliocostalis Lumborum pars Thoracis muscles were measured bilaterally. sEMG of the Anterior Deltoid muscle of the dominant arm was also measured. This RAM was used to induce an internal perturbation to the postural balance of subjects and is an often used task in the study of trunk motor control. Midway the RAM block, the participants got a short intermission of 90 seconds seated rest. Both conditions consisted of a warning cue (colored dot on a screen) followed by a go cue (arrow indicating either an upwards or downwards rapid arm movement) or a no-go cue ('STOP') and 12 seconds rest before the next trial. Harmless vibrotactile stimuli were always administered to the low back region during the appearance of the warning cue. During the C, a white warning cue was presented (safe cue), meaning that the RAM would never be accompanied by a painful electrocutaneous stimulus in that condition. During the F a safe (no threat) or a threatening warning cue could be presented (50-50%); in 25% of the trials after the threatening cue an electrocutaneous stimulus was given to the lower back region; the trials after the no threat cue were never accompanied with painful stimuli.

The intensity of the electrocutaneous stimulus was self-determined by participants through a staircase paradigm and was administered by a digitimer system.

At the beginning of each test day several questionnaires were also administered to control for psychological factors and physical activity, i.e. Central Sensitization Index (CSI), Hospital Anxiety and Depression Scale (HADS), Tampa Scale for Kinesiophobia (TSK), Pain Catastrophizing Scale (PCS), Pain Vigilance and Awareness Questionnaire (PVAQ), Roland-Morris Disability Questionnaire (RMDQ), International Physical Activity Questionnaire (IPAQ) and a general questionnaire regarding socio-demographic information and history of complaints. Furthermore, complaint specific questionnaires were also administered, but only for the clinical populations (RLBP and CLBP)

Statistical analysis will be performed to assess whether and to what extent both threat and LBP might influence motor control as measured with EMG during RAM. Furthermore, the effect of both on cortical movement preparation and somatosensory processing will also be assessed based on the EEG measurements.

ELIGIBILITY:
Healthy controls

Inclusion Criteria:

* Healthy adult subjects.

Exclusion Criteria:

* People with a history of pain or current pain
* severe pathologies
* traumata
* cardiorespiratory disorders
* neurological disorders
* vestibular disorders
* endocrinologic disorders
* psychiatric and cognitive disorders
* colour blindness
* sleeping disorders
* psychological disorders or major depressions
* major surgery to the spine or upper limbs
* clinically relevant malalignments and deformities
* malignancies
* substance abuse of alcohol or drugs
* consumption of analgesics without prescription 24 hours or with prescription two weeks before testing
* use of psychotropic medication
* extreme physical activities two days before testing
* professional athletes
* pregnant women or women < 1 year postnatally

RLBP

Inclusion Criteria:

* People with non-specific recurrent LBP for at least 2 episodes last year. (1 episode = >24h complaints; 2 episodes are separated by a painfree period of at least 1 month)

Exclusion Criteria:

* specific reason for LBP (e.g. herniation <2y, fracture, rheumatic disease,...)
* severe pathologies
* traumata
* cardiorespiratory disorders
* neurological disorders
* vestibular disorders
* endocrinologic disorders
* psychiatric and cognitive disorders
* colour blindness
* sleeping disorders
* psychological disorders or major depressions
* major surgery to the spine or upper limbs
* clinically relevant malalignments and deformities
* malignancies
* substance abuse of alcohol or drugs
* consumption of analgesics without prescription 24 hours or with prescription two weeks before testing
* use of psychotropic medication
* extreme physical activities two days before testing
* professional athletes
* pregnant women or women < 1 year postnatally

CLBP

Inclusion Criteria:

* People with non-specific chronic LBP for at least 3 days a week and this for at least 3 months on a row.

Exclusion Criteria:

* specific reason for LBP (e.g. herniation <2y, fracture, rheumatic disease,...)
* severe pathologies
* traumata
* cardiorespiratory disorders
* neurological disorders
* vestibular disorders
* endocrinologic disorders
* psychiatric and cognitive disorders
* colour blindness
* sleeping disorders
* psychological disorders or major depressions
* major surgery to the spine or upper limbs
* clinically relevant malalignments and deformities
* malignancies
* substance abuse of alcohol or drugs
* consumption of analgesics without prescription 24 hours or with prescription two weeks before testing
* use of psychotropic medication
* extreme physical activities two days before testing
* professional athletes
* pregnant women or women < 1 year postnatally

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Trunk muscle EMG latency | 2 hours
  Latency of the activation onset of the trunk muscles on EMG compared to prime mover onset (Anterior Deltoid) in milliseconds.
Contingent Negative Variation | 2 hours
  A cortical EEG-potential that reflects movement preparation in the timeframe between a warning cue and a go cue in Volt.
Somatosensory Evoked Potentials | 2 hours
  Cortical EEG-potentials that reflect the awareness and processing of somatosensory information, in this case vibrotactile stimuli on the lower back in Herz.

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain | Before, midway and after each RAM block, with a duration of 10 seconds. This in both test day 1 and 2, which are minimally separated by 5 days between test days.
  A self-reported rating by participants for experienced low back pain, which was assessed at baseline, midway the RAM block (during the 90s intermission) and after the RAM. Participants had to indicate on a horizontal axis of 10 cm how much LBP they experienced at that moment with at the left side of the axis (0) 'no pain all' and on the right side of the axis (10) 'maximal/worst pain ever experienced'. The numeric score (0-10) was calculated by the researcher and was not visible for participants.
Rating of Perceived Exertion/Borg | After each RAM block, with a duration of 5 seconds. This in both test day 1 and 2, which are minimally separated by 5 days between test days.
  A self-reported rating by participants for assessing how fatiguing the RAM was. This was assessed after the RAM task. This is a vertical scale ranging from 6 at the top (no exertion) to 20 at the bottom ('maximal exertion') of the scale. Participants saw both incremental numbers from 6-20 and descriptions at numbers 7 ('very very light'), 9 ('very light'), 11 ('reasonably light'), 13 ('quite heavy'), 15 ('heavy'), 17 ('very heavy'), 19 ('very very heavy'), 20 ('maximal exertion').
International Physical Activities Questionnaire | 15 minutes at the beginning of each of two test days, which are minimally separated by 5 days between test days.
  The IPAQ was administered before each test session to question participants about the physical activities they performed during the last 7 days. This in order to control for week-to-week differences in physical exertion levels and in order to compare physical activity between subjects. Based on these scores 3 levels of physical activity could be determined with level 1 (low), 2 (moderate) and 3 (high) physical activity. These levels are calculated based on the amount of hours low, moderate and high exerting activities had been performed the last 7 days.
General Questionnaire | 10 minutes at the beginning of test day 1
  Demographical and physical characteristics were questioned in a self-developed general questionnaire as well as educational/occupational levels, substance and medication use, general physical and mental health at the beginning of test day 1.
General Questionnaire - Short | 10 minutes at the beginning of test day 2
  Only a short part of the General Questionnaire was repeated at the start of test day two. Demographic, physical and educational/occupational information would not alter between 2 test days, so these sections were unnecessary to question again at test day 2. Therefore a shorter version with only questions about substance and medication use since the previous test day, general physical and mental health was administered on test day 2.
Hospital Anxiety and Depression Scale (HADS) | 7 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The HADS was administered before each test day in order to be able to assess feelings of anxiety and depression experienced during the last week. This without including physical aspects, but solely the mental aspects thereof. 14 items (7 for anxiety, 7 for depression) had to be answered on a 4-point Likert scale (0-3). A total score would then be calculated ranging from 0-7 (no depression/anxiety), over 8-10 (possible depression/anxiety), to 11-21 (likely depression/anxiety).
Pain Catastrophizing Scale (PCS) | 7 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The PCS is a self-assessment scale that gives a valid indication of the amount of catastrophizing in both clinical and non-clinical populations. Catastrophizing plays an important role in the experience and consequent handling of pain. 13 statements have to be scored on a 5-point scale ranging from 0 ('not at all applicable') to 4 ('always applicable'). Total scores (0-52) as well as subscales for rumination (4 items), magnification (3 items) and helplessness (6 items) can be calculated.
Tampa Scale for Kinesiophobia (TSK) | 8 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The TSK is a questionnaire that assesses pain-related fear during everyday movements, and is mostly used for CLBP and fibromyalgia patient groups. It consists out of 17 items that can be subdivided into pathological somatic focus (5 items) and activity avoidance (8 items) questions. All statements have to be scored on a 4-point score, ranging from 1 ('strongly disagree') to 4 ('strongly agree'). A total score is calculated after inversion of the individual scores of items 4, 8, 12 and 16. A total score, and subscores for pathological somatic focus (5-20), and activity avoidance (8-32) can be calculated.
Pain Vigilance and Awareness Questionnaire (PVAQ) | 8 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The PVAQ is a broad measure of attention to pain, which can be applied to various pain populations. It consists of 16 statements, and respondents have to indicate on a 6-point scale (0 = never, 6 = always) the extent to which these statements correspond to their behaviour in the last week.
Roland Morris Disability Questionnaire (RMDQ) | 10 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The RMDQ specifically measures the physical condition of people with low back pain complaints and the manner in which this interferes with daily activities. It consists out of 24 questions about activities that might be disturbed by LBP. Respondents have to answer 'yes' or 'no' on each question to, leading to a total score (0-24) that reflects the amount of disability experienced.
Central Sensitization Inventory (CSI) | 10 minutes at the beginning of test day 1 and 2, which are minimally separated by 5 days between test days.
  The CSI is a questionnaire that assesses to which extent several central sensitization related aspects are present in the respondents. Therefore, respondents are required to score 25 statements on a 5-point Likert scale ranging from 0 ('never') to 4 ('always'). Furthermore, previous diagnostics of 10 sensitization-related syndromes (like fibromyalgia) are also assessed. Total scores on the CSI are divided subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100) regarding presence of central sensitization aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, PT, PhD, Principal Investigator — University Ghent
Locations (1):
- Vakgroep REVAKI (Ghent University - Ghent University Hospital), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared after completion of the study.